CLINICAL TRIAL: NCT07365254
Title: Accurate Assessment and Intervention Research on Newborn Whole Genome Sequencing and Genetic Disease Risk(China Baby Omics)
Brief Title: Accurate Assessment and Intervention Research on Newborn Whole Genome Sequencing and Genetic Disease Risk
Status: Recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20250021-R
Record Dates: First submitted 2025-08-25; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-01

CONDITIONS: Genetic Disease
Keywords: Newborn; Multiomics
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, vaginal secretions, feces, amniotic cells, umbilical cord blood, pregnancy outcome (POC), placental tissue, or other tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Maternal and infant health is the foundation of public health, and its status directly reflects the overall health level of the population. With rapid socioeconomic development and increasingly severe environmental issues, health problems among women and children have become more widespread and diverse. In the new era, maternal and child health faces new challenges, with higher demands in areas such as reproductive health promotion, birth defect prevention, maternal and infant safety, and childhood disease prevention. Cohort studies, as an epidemiological research method for exploring disease etiology, involve recruiting participants before or during pregnancy and conducting follow-ups on pregnancy, childbirth, and maternal and child health outcomes after birth to identify various factors influencing diseases and health. Focusing on the early stages of life, this approach is an effective method for studying the associations between environmental, genetic, and behavioral risk factors during early life and embryonic development, fetal health, and infant health.

This project plans to conduct long-term follow-ups on couples and their offspring on a family basis, while collecting biological samples at multiple time points. A systematic multi-dimensional assessment, based on clinical information and multi-omics data from the enrolled population, will be used to infer the causes of reproductive and pregnancy-related diseases and developmental abnormalities, identify new biomarkers for pregnancy-related diseases, establish predictive models, and recognize risk factors in the early life of offspring, thereby providing guidance for the prevention and control of reproductive and developmental diseases.

DETAILED DESCRIPTION:
If the donor agrees to participate in this project, they will need to sign a written informed consent form, register for enrollment, and complete relevant questionnaires. During the project participation, they will be required to provide a small amount of biological samples within the specified timeframe. The biological samples provided by the donor will be used by the project's collaborating institutions in the hospital to conduct multi-omics experiments and analyses, including nucleic acid extraction, detection, database construction, and sequencing of biological samples such as peripheral blood, urine, and vaginal secretions. The clinical data of the donor will be stored in the hospital, and the gene, protein, metabolic, and vaginal microbiome-related detection data generated based on the samples will also be stored in the hospital. The use of samples is subject to strict review procedures to ensure the rationality and feasibility of scientific research, as well as compliance with laws, regulations, and ethical norms.

ELIGIBILITY:
Inclusion Criteria:

* Families with ongoing pregnancies (via assisted reproductive therap or natural conception) and newborn infants.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Families with ongoing pregnancies (via assisted reproductive therap or natural conception) and newborn infants.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Whole-genome sequencing data | After the completion of sample collection, an average of 1 year.
  Complete 30-40X whole-genome sequencing of the serum cfDNA sample according to the instructions of the DNBSEQ-T7RS High-throughput Sequencing Kit (FCL PE100) V2.0, and perform bioinformatics analysis of the sequencing data.
Concentration of metabolite | After the completion of sample collection, an average of 1 year.
  The concentration of each metabolite was analyzed and calculated using the automated targeted metabolic absolute quantification software HMQuant, independently developed by BGI.
Construction and sequencing of cfRNA from maternal peripheral blood | After the completion of sample collection, an average of 1 year.
  The library construction and quality control were performed according to the BGI PALM-seq library construction method, followed by cfRNA sequencing. The PALM-seq sequencing bioinformati
Whole-genome DNA methylation data | After the completion of sample collection, an average of 1 year.
  Combining bisulfite treatment with high-throughput sequencing technology enables the efficient and accurate mapping of whole-genome DNA methylation profiles, making it a crucial tool for epigenomics research. Based on the domestically developed DNBSEQTM sequencing technology, BGI has independently developed a novel library preparation method utilizing double-strand cyclization. This approach effectively addresses the base bias issue present in traditional methylation sequencing, allowing for rapid and efficient acquisition of authentic methylation level data.
Protein expression differences and functional analysis | After the completion of sample collection, an average of 1 year.
  Sample protein preparation: Samples were taken from -80°C, and 50 μL of each sample was treated with urea, dithiothreitol, and iodoacetamide for reduction and alkylation. Solid-phase extraction plates were used to remove high-abundance proteins, followed by the addition of trypsin for enzymatic hydrolysis. Liquid chromatography-mass spectrometry detection: After enzymatic hydrolysis, the peptides were analyzed using nanoflow-high-performance liquid chromatography-high-resolution mass spectrometry (Lumos, Thermo) in DIA (data-independent acquisition) mode for data acquisition. Data analysis: DIA-NN software was used to identify and quantify proteins from the DIA data.
The metagenomic data | After the completion of sample collection, an average of 1 year.
  Vaginal secretion DNA extraction and library sequencing: Magpure Stoll DNA KF kit was used to extract DNA from vaginal secretions; Construct a metagenomic library using the MGIEasy universal DNA library preparation kit; Use Agilent 2100 Bioanalyzer to detect the fragment range and concentration of the library. Qualified libraries were sequenced using the T1 sequencing platform according to the DNBSEQ-T7RS high-throughput sequencing kit instructions. Bioinformatics analysis of metagenomic sequencing data: The metagenomic data is first subjected to quality control of the original sequences using Trimomatic software, and then contaminated sequences are removed from the processed data using fastq_streen software, including host sequences and phix library contamination; Afterwards, the BWA aligner was used for comparison, and the human genome fragments were first removed. The microbial species composition and relative abundance were evaluated using the Metaphlan2 software.

CONTACTS AND LOCATIONS:
Overall Officials: Hefeng Huang, Study Chair — Women's Hospital School Of Medicine Zhejiang University; Dan Zhang, Study Chair — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No